CLINICAL TRIAL: NCT02294461
Title: Asian Multinational Phase 3, Randomized, Double-Blind, Placebo-Controlled Efficacy and Safety Study of Oral Enzalutamide in Chemotherapy Naïve Subjects With Progressive Metastatic Prostate Cancer Who Have Failed Androgen Deprivation Therapy
Brief Title: An Asian Study to Evaluate Efficacy and Safety of Oral Enzalutamide in Progressive Metastatic Prostate Cancer Participants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 9785-CL-0232; CTR20140131 (Registry Identifier: ChinaDrugTrials.org.cn)
Record Dates: First submitted 2014-11-13; First posted 2014-11-19 (Estimated); Results first posted 2017-04-12 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Progressive Metastatic Prostate Cancer
Keywords: Enzalutamide; Androgen receptor; Prostate cancer; Xtandi
MeSH Terms: conditions — Bulbo-Spinal Atrophy, X-Linked; Prostatic Neoplasms | interventions — enzalutamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Enzalutamide (Experimental): Participants received 160 mg of enzalutamide orally once a day during double blind period until Prostate-Specific Antigen (PSA) progression and radiographic disease progression were centrally confirmed and 1 of the following 2 events became applicable to the participants: (1) initiation of cytotoxic chemotherapy or (2) initiation of an investigational agent for treatment of prostate cancer. Eligible participants who received enzalutamide during double blind and who provided consent to take part in open-label period continued to receive 160 mg of enzalutamide in open-label period orally once a day until PSA progression and radiographic disease progression were centrally confirmed and 1 of the following 2 events became applicable to the participants: (1) initiation of cytotoxic chemotherapy or (2) initiation of an investigational agent for treatment of prostate cancer.
  Interventions: Drug: Enzalutamide
- Placebo (Experimental): Participants received enzalutamide matching placebo orally once a day during double-blind period until PSA progression and radiographic disease progression were centrally confirmed and 1 of the following 2 events became applicable to the participants: (1) initiation of cytotoxic chemotherapy or (2) initiation of an investigational agent for treatment of prostate cancer.
  Interventions: Drug: Placebo
- Placebo followed by Enzalutamide (Experimental): Eligible participants who received enzalutamide matching placebo during double-blind period and who provided consent to take part in open-label period, received 160 mg of enzalutamide orally once a day during open-label period until PSA progression and radiographic disease progression were centrally confirmed and 1 of the following 2 events became applicable to the participants: (1) initiation of cytotoxic chemotherapy or (2) initiation of an investigational agent for treatment of prostate cancer.
  Interventions: Drug: Enzalutamide

INTERVENTIONS:
Drug: Enzalutamide — Oral
  Other Names: Xtandi; MDV3100
  Arms: Enzalutamide; Placebo followed by Enzalutamide
Drug: Placebo — Oral
  Arms: Placebo

SUMMARY:
Purpose of the study was to assess the effect of enzalutamide on time to Prostate Specific Antigen (PSA) progression as compared to placebo in chemotherapy naïve participants with progressive metastatic prostate cancer who have failed androgen deprivation therapy.

DETAILED DESCRIPTION:
The study was a multinational Phase 3, randomized, double-blind, placebo-controlled efficacy and safety study of oral enzalutamide (formerly MDV3100) in asymptomatic or mildly symptomatic participants with progressive metastatic prostate cancer who have disease progression despite androgen deprivation therapy. In order to join the study, participants could not have been previously treated with cytotoxic chemotherapy. Approximately 30 Chinese participants were allocated to the pharmacokinetic (PK) cohort. Participants in the PK cohort were required to be hospitalized from Day 1 before the randomization date to at least the completion of all the assessments planned on Day 3. All participants in the PK cohort underwent blood sampling for the PK analysis. Data reported in the results section was based on data cutoff dates of 20 Sept 2015 for efficacy and safety data and 20 Jan 2016 for PK outcome measures. The study completed double-blind period and is now in the open-label period.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation or small cell features
* Ongoing androgen deprivation therapy with a GnRH analogue or bilateral orchiectomy
* Progressive disease despite androgen deprivation therapy as defined by rising PSA levels or progressive soft tissue or bone disease
* No prior treatment with cytotoxic chemotherapy
* Asymptomatic or mildly symptomatic from prostate cancer

Exclusion Criteria:

* Severe concurrent disease, infection, or co-morbidity that, in the judgment of the Investigator, would make the patient inappropriate for enrollment
* Known or suspected brain metastasis or active leptomeningeal disease
* History of another malignancy within the previous 5 years other than curatively treated non-melanomatous skin cancer
* History of seizure including febrile seizure or any condition that may predispose to seizure (e.g., prior stroke, brain arteriovenous malformation, head trauma with loss of consciousness requiring hospitalization).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 395 (Actual)
Dates: Start 2014-04-23 (Actual); Primary Completion 2015-09-20 (Actual); Study Completion 2024-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Astellas Pharma Inc
Locations (47):
- China (22):
  - CN00103, Beijing
  - CN00104, Beijing
  - CN00106, Beijing
  - CN00111, Beijing
  - CN00112, Beijing
  - CN00114, Beijing
  - CN00115, Beijing
  - CN00127, Beijing
  - CN00121, Changsha
  - CN00107, Hangzhou
  - CN00110, Nanjing
  - CN00117, Nanjing
  - CN00102, Shanghai
  - CN00105, Shanghai
  - CN00108, Shanghai
  - CN00113, Shanghai
  - CN00126, Shanghai
  - CN00119, Suzhou
  - CN00125, Tianjin
  - CN00118, Wenzhou
  - CN00109, Wuhan
  - CN00124, Xi'an
- HK00402, Hong Kong, Hong Kong
- South Korea (15):
  - KR00214, Anyang
  - KR00205, Busan
  - KR00207, Busan
  - KR00212, Cheongju-si
  - KR00203, Daegu
  - KR00213, Daejeon
  - KR00201, Incheon
  - KR00202, Seongnam-si
  - KR00204, Seoul
  - KR00206, Seoul
  - KR00208, Seoul
  - KR00209, Seoul
  - KR00210, Seoul
  - KR00211, Seoul
  - KR00215, Seoul
- Taiwan (9):
  - TW00309, Kaohsiung City
  - TW00302, Taichung
  - TW00303, Taichung
  - TW00307, Tainan
  - TW00308, Tainan
  - TW00301, Taipei
  - TW00304, Taipei
  - TW00306, Taipei
  - TW00305, Taoyuan

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Pu YS, Ahn H, Han W, Huang SP, Wu HC, Ma L, Yamada S, Suga K, Xie LP. Enzalutamide in Chemotherapy-Naive Metastatic Castration-Resistant Prostate Cancer: An Asian Multiregional, Randomized Study. Adv Ther. 2022 Jun;39(6):2641-2656. doi: 10.1007/s12325-022-02140-2. Epub 2022 Apr 10. PMID 35397772
- See also: Link to results and other applicable study documents on the Astellas Clinical Trials website. — https://www.clinicaltrials.astellas.com/study/9785-CL-0232
- See also: Link to plain language summary of the study on the Trial Results Summaries website. — https://www.trialsummaries.com/Study/StudyDetails?id=14501&tenant=MT_AST_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study population consisted of men with asymptomatic or mildly symptomatic progressive metastatic prostate cancer, who had failed androgen deprivation therapy, and have not been treated with cytotoxic chemotherapy. Participants from 46 study sites in 4 countries (China, Korea, Taiwan and Hong Kong) were randomized for the study.
Pre-assignment Details: Participants who met inclusion criteria and none of the exclusion criteria were enrolled in the study.
Groups:
- Enzalutamide: Participants received 160 milligrams (mg) of enzalutamide orally once a day during double blind period until Prostate-Specific Antigen (PSA) progression and radiographic disease progression were centrally confirmed and 1 of the following 2 events became applicable to the participants: (1) initiation of cytotoxic chemotherapy or (2) initiation of an investigational agent for treatment of prostate cancer (up to 29.4 months). Eligible participants who received enzalutamide during double blind and who provided consent to take part in open-label period continued to receive 160 mg of enzalutamide in open-label period orally once a day until PSA progression and radiographic disease progression were centrally confirmed and 1 of the following 2 events became applicable to the participants: (1) initiation of cytotoxic chemotherapy or (2) initiation of an investigational agent for treatment of prostate cancer (up to 54.3 months).
- Placebo: Participants received enzalutamide matching placebo orally once a day during double-blind period until PSA progression and radiographic disease progression were centrally confirmed and 1 of the following 2 events became applicable to the participants: (1) initiation of cytotoxic chemotherapy or (2) initiation of an investigational agent for treatment of prostate cancer (up to 18.6 months).
- Placebo Patients Crossover to Enzalutamide 160 mg: Eligible participants who received enzalutamide matching placebo during Double Blind period and who provided consent to take part in Open label period, received 160 mg of enzalutamide orally once a day during open-label period until PSA progression and radiographic disease progression were centrally confirmed and 1 of the following 2 events became applicable to the participants: (1) initiation of cytotoxic chemotherapy or (2) initiation of an investigational agent for treatment of prostate cancer (up to 53.8 months).
Period: Double-blind Period (up to 29.4 Months)
Arm/Group | Enzalutamide | Placebo | Placebo Patients Crossover to Enzalutamide 160 mg
Started | 202 | 193 | 0
Treated/Received Study Drug | 202 | 193 | 0
Completed | 84 | 1 | 0
Not Completed | 118 | 192 | 0
Not completed — Death | 6 | 4 | 0
Not completed — Miscellaneous | 30 | 66 | 0
Not completed — Withdrawal by Subject | 27 | 54 | 0
Not completed — Protocol Deviation | 0 | 2 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Progressive Disease | 38 | 51 | 0
Not completed — Adverse Event | 16 | 15 | 0
Period: Open-label Period (up to 54.3 Months)
Arm/Group | Enzalutamide | Placebo | Placebo Patients Crossover to Enzalutamide 160 mg
Started | 85 (Eligible participants who provided consent took part in open-label period.) | 0 (Eligible participants who provided consent took part in open-label period.) | 51 (Eligible participants who provided consent took part in open-label period.)
Completed | 0 | 0 | 0
Not Completed | 85 | 0 | 51
Not completed — Miscellaneous | 28 | 0 | 16
Not completed — Withdrawal by Subject | 19 | 0 | 10
Not completed — Protocol Deviation | 2 | 0 | 0
Not completed — Lost to Follow-up | 4 | 0 | 2
Not completed — Progressive Disease | 20 | 0 | 12
Not completed — Death | 6 | 0 | 5
Not completed — Adverse Event | 6 | 0 | 6

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population consisted of all randomized participants in the study.
Groups:
- Enzalutamide: Participants received 160 mg of enzalutamide orally once a day during double blind period until PSA progression and radiographic disease progression were centrally confirmed and 1 of the following 2 events became applicable to the participants: (1) initiation of cytotoxic chemotherapy or (2) initiation of an investigational agent for treatment of prostate cancer (up to 29.4 months). Eligible participants who received enzalutamide during double blind and who provided consent to take part in open-label period continued to receive 160 mg of enzalutamide in open-label period orally once a day until PSA progression and radiographic disease progression were centrally confirmed and 1 of the following 2 events became applicable to the participants: (1) initiation of cytotoxic chemotherapy or (2) initiation of an investigational agent for treatment of prostate cancer (up to 54.3 months).
- Placebo: Participants received enzalutamide matching placebo orally once a day during double-blind period until PSA progression and radiographic disease progression were centrally confirmed and 1 of the following 2 events became applicable to the participants: (1) initiation of cytotoxic chemotherapy or (2) initiation of an investigational agent for treatment of prostate cancer (up to 18.6 months). Eligible participants who received enzalutamide matching placebo during double-blind period and who provided consent to take part in open-label period, received 160 mg of enzalutamide orally once a day during open-label period until PSA progression and radiographic disease progression were centrally confirmed and 1 of the following 2 events became applicable to the participants: (1) initiation of cytotoxic chemotherapy or (2) initiation of an investigational agent for treatment of prostate cancer (up to 53.8 months).
- Total: Total of all reporting groups
Arm/Group | Enzalutamide | Placebo | Total
Number analyzed (Participants) | 202 | 193 | 395
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.6 (8.1) | 71 (8.7) | 71.3 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 202 | 193 | 395
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 202 | 193 | 395
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Time to Prostate-specific Antigen (PSA) Progression
Description: The time to Prostate Specific Antigen (PSA) progression was defined as the time from randomization to the PSA progression. The PSA progression was defined according to the consensus guidelines of Prostate Cancer Clinical Trials Working Group 2 (PCWG2).For participants with PSA decline at Week 13, the PSA progression date was defined as a ≥ 25% increase and an absolute increase of ≥ 2 ng/mL above the nadir, which would be confirmed by a second consecutive value obtained 3 or more weeks later. For participants with no PSA decline at Week 13, the PSA progression date was defined as the date when a ≥ 25% increase and an absolute increase of ≥ 2 ng/mL above the baseline was documented, which was confirmed by a second consecutive value 3 or more weeks later. Time to PSA progression was estimated using the Kaplan-Meier method. Participants without confirmed PSA progression were censored.
Time Frame: From the date of randomization to PSA progression median follow-up time is 6.47 months for enzalutamide and 2.99 months for placebo
Population: ITT population with available data.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Enzalutamide | Placebo
Number analyzed (Participants) | 198 | 190
Months | 8.31 [5.72 to 10.25] | 2.86 [2.83 to 4.63]
Statistical Analysis 1: Comparison: Enzalutamide vs Placebo; P-value is based on an unstratified log-rank test. Hazard ratio calculated using unstratified Cox Proportional Hazards model with treatment as the only covariate for enzalutamide group versus placebo group; Test type: Superiority or Other; p < 0.0001, Hazard Ratio; Unstratified Cox Proportional Hazards = 0.38, 95% CI 2-sided [0.27 to 0.52]

2. Secondary Outcome: Duration of Overall Survival
Description: Duration of overall survival was defined as the time from the randomization to deaths from any cause. For participants who were alive at the time of the data analysis, overall survival time was censored to the last know date the participants were known to be alive.
Time Frame: From the date of randomization to deaths from any cause median follow-up time is 42.32 months for enzalutamide and 26.81 months for placebo
Population: ITT population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Enzalutamide | Placebo
Number analyzed (Participants) | 202 | 193
Months | 39.06 [29.24 to 57.63] | 27.10 [21.88 to 37.82]
Statistical Analysis 1: Comparison: Enzalutamide vs Placebo; Participants who were not known to have had died at the analysis date were censored at date last known alive. Hazard ratio calculated using unstratified Cox Proportional Hazards model with treatment as the only covariate for enzalutamide group versus placebo group; Test type: Superiority or Other; p = 0.0208, Unstratified log-rank test — P-value is based on an unstratified log-rank test; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.51 to 0.95]

3. Secondary Outcome: Duration of Radiographic Progression-free Survival (rPFS) Based on Independent Central Review Facility Assessment
Description: Duration of Radiographic Progression-free Survival (rPFS) was defined as the time from randomization to the rPFS event (deaths from any cause and radiographic disease progression). Radiographic disease progression is defined by RECIST 1.1 for soft tissue disease, or PCWG2 for bone lesions. If a participant met the criteria for more than 1 censoring rule, they were censored with the earliest censoring date. The radiographic progression date was the first date when progression definition was met, not confirmed.
Time Frame: From the date of randomization to the rPFS event (deaths from any cause and radiographic disease progression) median follow-up time is 5.55 months for enzalutamide and 3.71 months for placebo
Population: ITT population with available data.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Enzalutamide | Placebo
Number analyzed (Participants) | 198 | 190
Months | NA [10.97 to NA] — Could not be estimated due to the low number of events | 5.29 [3.61 to 11.33]
Statistical Analysis 1: Comparison: Enzalutamide vs Placebo; Participants who were not known to have had an rPFS event were censored at the date of the last assessment showing no objective evidence of rPFS prior to scan modality change, new antineoplastic treatment, initiation of radiation therapy for prostate cancer, skeletal-related event (SRE) and 2 or more consecutive missed tumor assessments. Hazard ratio calculated using unstratified Cox Proportional Hazards model with treatment as the only covariate for enzalutamide; Test type: Superiority or Other; p < 0.0001, Unstratified log-rank test — P-value is based on an unstratified log-rank test; Hazard Ratio (HR) = 0.31, 95% CI [0.20 to 0.46]

4. Secondary Outcome: Time to First Skeletal-Related Event
Description: Time to first skeletal-related event (SRE) was defined as the time from randomization to the first skeletal-related event, defined as radiation therapy or surgery to bone, pathologic bone fracture, spinal cord compression, or change of anti-neoplastic therapy to treat bone pain. Participants who have not had a SRE at the time of the analysis were censored at their last assessment indicating no evidence of SRE.
Time Frame: From the date of randomization to the first skeletal-related event median follow-up time is 7.39 months for enzalutamide and 5.29 months for placebo
Population: ITT population with available data.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Enzalutamide | Placebo
Number analyzed (Participants) | 198 | 190
Months | NA [NA to NA] — Could not be estimated due to the low number of events | NA [NA to NA] — Could not be estimated due to the low number of events
Statistical Analysis 1: Comparison: Enzalutamide vs Placebo; Participants who did not have an SRE were censored at the date of the last assessment indicating no evidence of SRE. Hazard ratio calculated using unstratified Cox Proportional Hazards model with treatment as the only covariate for enzalutamide group versus placebo group; Test type: Superiority or Other; p = 0.2501, Unstratified log-rank test — P-value was based on an unstratified log-rank test; Hazard Ratio (HR) = 0.56, 95% CI 2-sided [0.21 to 1.52]

5. Secondary Outcome: Time to Initiation of Cytotoxic Chemotherapy
Description: Time to initiation of cytotoxic chemotherapy was defined as the time from randomization to initiation of cytotoxic chemotherapy. It included only therapies for prostate cancer. When multiple cytotoxic chemotherapies were initiated, the first chemotherapy was used to determine the time to event. Participants who did not start cytotoxic chemotherapy at the time of analysis data cutoff were censored at the date of their last assessment indicating no evidence of cytotoxic chemotherapy usage.
Time Frame: From the date of randomization to initiation of cytotoxic chemotherapy median follow-up time is 7.39 months for enzalutamide and 5.19 months for placebo
Population: ITT population with available data.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Enzalutamide | Placebo
Number analyzed (Participants) | 198 | 190
Months | NA [NA to NA] — Could not be estimated due to the low number of events | 13.93 [NA to NA] — Could not be estimated due to the low number of events
Statistical Analysis 1: Comparison: Enzalutamide vs Placebo; Participants who did not start cytotoxic chemotherapy were censored at the date of the last assessment indicating no evidence of cytotoxic chemotherapy usage. Hazard ratio calculated using unstratified Cox Proportional Hazards model with treatment as the only covariate for enzalutamide group versus placebo group; Test type: Superiority or Other; p = 0.0020, Unstratified log-rank test — P-value is based on an unstratified log-rank test; Hazard Ratio (HR) = 0.28, 95% CI [0.12 to 0.66]

6. Secondary Outcome: Number of Participants With Confirmed Best PSA Response (≥50% Decrease From Baseline)
Description: Best PSA response was defined as as ≥50% reductions in PSA level from baseline to the lowest post-baseline PSA result as determined by the central laboratory, with a consecutive assessment conducted at least 3 weeks later to confirm the PSA response. Only participants who had both baseline and post-baseline assessments were included in the analysis.
Time Frame: From baseline to the lowest post-baseline PSA result median treatment duration is 6.60 months for enzalutamide and 3.70 months for placebo
Population: ITT population with available data.
Measure: Number; unit: Participants
Arm/Group | Enzalutamide | Placebo
Number analyzed (Participants) | 182 | 148
Participants | 120 | 15
Statistical Analysis 1: Comparison: Enzalutamide vs Placebo; Test type: Superiority or Other; p < 0.0001, Unstratified Cochran-Mantel-Haenszel % — P-value is based on unstratified Cochran-Mantel-Haenszel mean score test; Difference of response rate = 55.8, 95% CI 2-sided [47.4 to 64.2]

7. Secondary Outcome: Best Overall Soft Tissue Response
Description: Participants with measurable soft tissue disease at screening visit (i.e., at least one target lesion per Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1) who have an objective response (complete response (CR) or partial response (PR)) during the study were included in the best overall soft tissue response assessment. The best overall soft tissue response was based on the investigator assessment using RECIST 1.1. CR was defined as complete resolution of all attributable clinical symptoms and physical findings. PR was defined as partial resolution of at Least some of the clinical symptoms and physical findings.
Time Frame: From the date of randomization median treatment duration is 6.60 months for enzalutamide and 3.70 months for placebo
Population: ITT population with available data.
Measure: Number; unit: Participants
Arm/Group | Enzalutamide | Placebo
Number analyzed (Participants) | 65 | 60
Participants | 18 | 1
Statistical Analysis 1: Comparison: Enzalutamide vs Placebo; When deriving the response category, it was based on the target, non-target and new lesions without confirming CR, PR, and Progressive disease (PD). Participants with no post baseline assessment were included in the category of Nonevaluable (NE). The best overall soft tissue objective response was defined as PR or CR based on the investigator assessments of target, non-target and new lesions while on the study treatment; Test type: Superiority or Other; p < 0.0001, Unstratified Cochran-Mantel-Haenszel — P-value is based on unstratified Cochran-Mantel-Haenszel mean score test; Difference in objective response rate = 26.0, 95% CI 2-sided [14.7 to 37.4]

8. Secondary Outcome: Time to Maximum Concentration (Tmax) of Enzalutamide, M1,M2 and Enzalutamide Plus M2
Time Frame: From the date of randomization, Single Dosing Day 1 and Multiple Dosing Day 85
Population: The Pharmacokinetic Analysis Set (PKAS) population consisted of all participants who received at least 1 dose of study drug and who provided blood samples for drug concentrations at at least 1 time point.
Measure: Median (Full Range); unit: hour
Groups:
- M1- Carboxylic Acid Metabolite: Inactive metabolite
- M2- N-Desmethyl Enzalutamide: N-desmethyl enzalutamide (active metabolite)
- Enzalutamide Plus M2: Active metabolite
Arm/Group | Enzalutamide | M1- Carboxylic Acid Metabolite | M2- N-Desmethyl Enzalutamide | Enzalutamide Plus M2
Number analyzed (Participants) | 12 | 12 | 12 | 12
hour
  Day 1 | 0.975 [0.500 to 6.05] | 24.0 [0.550 to 24.9] | 24.0 [0.550 to 24.9] | 0.975 [0.500 to 24.0]
  Day 85: number analyzed (Participants) | 11 | 11 | 11 | 11
  Day 85 | 1.00 [0 to 2.00] | 1.02 [0.217 to 24.1] | 0 [0 to 23.8] | 0.250 [0 to 23.8]

9. Secondary Outcome: Maximum Observed Plasma Concentration During the First 24 Hours After Dosing (Cmax) Enzalutamide, M1,M2 and Enzalutamide Plus M2
Time Frame: From the date of randomization, Single Dosing Day 1 and Multiple Dosing Day 85
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: micrograms/milliliter (μg/mL)
Arm/Group | Enzalutamide | M1- Carboxylic Acid Metabolite | M2- N-Desmethyl Enzalutamide | Enzalutamide Plus M2
Number analyzed (Participants) | 12 | 12 | 12 | 12
micrograms/milliliter (μg/mL)
  Day 1 | 3.92 (1.37) | 0.112 (0.0794) | 0.175 (0.0921) | 3.94 (1.34)
  Day 85: number analyzed (Participants) | 11 | 11 | 11 | 11
  Day 85 | 20.0 (3.22) | 14.0 (23.5) | 15.2 (3.44) | 34.2 (4.98)

10. Secondary Outcome: AUC From the Time of Dosing to 24 h After Dosing (AUC24h) Enzalutamide, M1,M2 and Enzalutamide Plus M2
Time Frame: From the date of randomization, Single Dosing Day 1 and Multiple Dosing Day 85
Population: The Pharmacokinetic Analysis Set (PKAS) population consisted of all participants who received at least 1 dose of study drug and who provided blood samples for drug concentrations at at least 1 time point. Number of participants analyzed is the number of participants with available data at this time point.
Measure: Mean (Standard Deviation); unit: μg*h/mL
Arm/Group | Enzalutamide | M1- Carboxylic Acid Metabolite | M2- N-Desmethyl Enzalutamide | Enzalutamide Plus M2
Number analyzed (Participants) | 12 | 12 | 12 | 12
μg*h/mL | 43.1 (9.64) | 1.81 (0.972) | 2.17 (1.30) | 45.3 (10.1)

11. Secondary Outcome: Concentration 24 h After Dosing (C24h) Enzalutamide, M1,M2 and Enzalutamide Plus M2
Description: N is the number of participants with available data at this time point.
Time Frame: From the date of randomization, Single Dosing Day 1 and Multiple Dosing Day 85
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Enzalutamide | M1- Carboxylic Acid Metabolite | M2- N-Desmethyl Enzalutamide | Enzalutamide Plus M2
Number analyzed (Participants) | 12 | 12 | 12 | 12
μg/mL
  Day 1 | 1.65 (0.343) | 0.111 (0.0801) | 0.164 (0.0942) | 1.82 (0.363)
  Day 85: number analyzed (Participants) | 10 | 10 | 10 | 10
  Day 85 | 17.6 (3.09) | 6.09 (3.07) | 13.7 (2.91) | 31.2 (4.00)

12. Secondary Outcome: Observed Plasma Concentration in Predose Samples Obtained During Multiple-dose Administration of Minimum Concentration (Plasma Concentration at Pre Dose) (Cmin) Enzalutamide, M1,M2 and Enzalutamide Plus M2
Description: N is the number of participants with available data at this time point.
Time Frame: From the date of randomization up to Days 2, 3, 8, 22, 29, 43, 57, 85, 86, 113, 141 and 169
Population: The Pharmacokinetic Analysis Set (PKAS) population consisted of all participants who received at least 1 dose of study drug and who provided blood samples for drug concentrations at least 1 time point.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Enzalutamide | M1- Carboxylic Acid Metabolite | M2- N-Desmethyl Enzalutamide | Enzalutamide Plus M2
Number analyzed (Participants) | 12 | 12 | 12 | 12
μg/mL
  Day 2 predose | 1.65 (0.343) | 0.111 (0.0801) | 0.164 (0.0942) | 1.82 (0.363)
  Day 3 predose | 3.29 (1.16) | 0.302 (0.256) | 0.367 (0.188) | 3.66 (1.24)
  Day 8 predose | 9.39 (2.07) | 1.21 (0.923) | 1.94 (0.983) | 11.3 (2.62)
  Day 22 predose: number analyzed (Participants) | 11 | 11 | 11 | 11
  Day 22 predose | 17.6 (2.37) | 6.09 (8.26) | 8.34 (2.74) | 25.9 (3.25)
  Day 29 predose | 19.6 (4.00) | 8.16 (12.5) | 10.9 (3.72) | 30.5 (5.47)
  Day 43 predose: number analyzed (Participants) | 11 | 11 | 11 | 11
  Day 43 predose | 17.0 (4.13) | 12.5 (22.1) | 14.0 (3.99) | 31.0 (5.82)
  Day 57 predose: number analyzed (Participants) | 11 | 11 | 11 | 11
  Day 57 predose | 17.8 (3.09) | 18.4 (28.2) | 14.7 (3.88) | 32.5 (4.57)
  Day 85 predose: number analyzed (Participants) | 11 | 11 | 11 | 11
  Day 85 predose | 17.9 (3.19) | 6.33 (2.95) | 14.9 (3.67) | 32.8 (5.10)
  Day 86 predose: number analyzed (Participants) | 10 | 10 | 10 | 10
  Day 86 predose | 17.6 (3.09) | 6.09 (3.07) | 13.7 (2.91) | 31.2 (4.00)
  Day 113 predose: number analyzed (Participants) | 7 | 7 | 7 | 7
  Day 113 predose | 17.5 (4.14) | 17.5 (33.1) | 15.0 (3.21) | 32.5 (3.72)
  Day 141 predose: number analyzed (Participants) | 6 | 6 | 6 | 6
  Day 141 predose | 17.3 (3.73) | 5.52 (2.10) | 14.3 (3.90) | 31.6 (4.70)
  Day 169 predose: number analyzed (Participants) | 4 | 4 | 4 | 4
  Day 169 predose | 17.2 (5.55) | 5.09 (2.27) | 14.0 (4.80) | 31.2 (5.02)

13. Secondary Outcome: Apparent Total Systemic Clearance After Multiple Dosing (CL/F) Enzalutamide, M1,M2 and Enzalutamide Plus M2 (For Unchanged Enzalutamide Only)
Time Frame: From the date of randomization up to Multiple Dosing Day 85
Population: as for outcome 8
Measure: Mean (Standard Error); unit: L/h
Groups:
- M2- N-Desmethyl Enzalutamide; Enzalutamide Plus M2: Active metabolite.
Arm/Group | Enzalutamide | M1- Carboxylic Acid Metabolite | M2- N-Desmethyl Enzalutamide | Enzalutamide Plus M2
Number analyzed (Participants) | 10 | 10 | 10 | 10
L/h | 0.387 (0.0774) | NA (NA) — Metabolite dose was unknown. | NA (NA) — Metabolite dose was unknown. | NA (NA) — Metabolite dose was unknown.

14. Secondary Outcome: Peak-Trough Ratio (PTR) Enzalutamide, M1,M2 and Enzalutamide Plus M2
Time Frame: From the date of randomization up to Multiple Dosing Day 85
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Enzalutamide | M1- Carboxylic Acid Metabolite | M2- N-Desmethyl Enzalutamide | Enzalutamide Plus M2
Number analyzed (Participants) | 10 | 10 | 10 | 10
Ratio | 1.15 (0.110) | 1.19 (0.364) | 1.09 (0.0897) | 1.08 (0.0581)

15. Secondary Outcome: AUC From the Time of Dosing to the Start of the Next Dosing Interval (AUCtau) Enzalutamide, M1,M2 and Enzalutamide Plus M2
Time Frame: From the date of randomization up to Multiple Dosing Day 85
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: μg*h/mL
Arm/Group | Enzalutamide | M1- Carboxylic Acid Metabolite | M2- N-Desmethyl Enzalutamide | Enzalutamide Plus M2
Number analyzed (Participants) | 10 | 10 | 10 | 10
μg*h/mL | 427 (79.8) | 149 (74.1) | 308 (68.2) | 735 (109)

16. Secondary Outcome: Number of Participants With Adverse Events (AE)
Description: An AE was defined as any untoward medical occurrence, temporally associated with use of medicinal product, whether considered related to medicinal product. AE could therefore be any unfavorable & unintended sign, symptom, or disease temporally associated with use of a medicinal product. An AE was considered serious if, results in death; is life-threatening; results in persistent disability; results in congenital anomaly; requires inpatient hospitalization; or leads to prolongation of hospitalization; other medically important events. TEAE was defined as AE occurring from time of study drug administration on Day 1 until follow-up visit (28 days after last dose, or one day before date of initiation of cytotoxic chemotherapy or an investigational agent, whichever comes first). AEs were graded using National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.03, where Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Life-threatening; Grade 5 = Fatal.
Time Frame: From first dose on Day 1 until 28 days after the last dose of study drug, or one day before the date of initiation of cytotoxic chemotherapy or an investigational agent for treatment of prostate cancer, whichever comes first, up to 123 months and 24 days
Population: Safety Analysis Set consisted of all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: Participants
Groups:
- Enzalutamide: Participants received 160 mg of enzalutamide orally once a day during double blind period until PSA progression and radiographic disease progression were centrally confirmed and 1 of the following 2 events became applicable to the participants: (1) initiation of cytotoxic chemotherapy or (2) initiation of an investigational agent for treatment of prostate cancer (up to 29.4 months). Eligible participants who received enzalutamide during double blind and who provided consent to take part in open-label period continued to receive 160 mg of enzalutamide in open-label period orally once a day until PSA progression and radiographic disease progression were centrally confirmed and 1 of the following 2 events became applicable to the participants: (1) initiation of cytotoxic chemotherapy or (2) initiation of an investigational agent for treatment of prostate cancer (up to 54.3 months). This arm represents both double blind and open-label period.
- Placebo: Participants received enzalutamide matching placebo orally once a day during double-blind period until PSA progression and radiographic disease progression were centrally confirmed and 1 of the following 2 events became applicable to the participants: (1) initiation of cytotoxic chemotherapy or (2) initiation of an investigational agent for treatment of prostate cancer (up to 18.6 months). This arm represents only double blind period.
- Placebo Followed by Enzalutamide: Eligible participants who received enzalutamide matching placebo during double-blind period and who provided consent to take part in open-label period, received 160 mg of enzalutamide orally once a day during open-label period until PSA progression and radiographic disease progression were centrally confirmed and 1 of the following 2 events became applicable to the participants: (1) initiation of cytotoxic chemotherapy or (2) initiation of an investigational agent for treatment of prostate cancer (up to 53.8 months). This arm represents only open-label period.
Arm/Group | Enzalutamide | Placebo | Placebo Followed by Enzalutamide
Number analyzed (Participants) | 202 | 193 | 51
Participants
  Treatment Emergent Adverse Events (TEAEs) | 190 | 166 | 47
  Grade 3 or Higher TEAE | 98 | 66 | 28
  TEAE Leading to Death | 24 | 7 | 7
  Serious TEAE | 87 | 57 | 24
  TEAE That Was Primary Reason for Treatment Discontinuation | 32 | 33 | 7
  TEAE Leading to Study Drug Discontinuation | 49 | 42 | 12
  TEAE Leading to Dose Reduction of Study Drug | 4 | 3 | 2
  TEAE Leading to Dose Interruption of Study Drug | 28 | 16 | 7
  TEAE Related to Study Drug | 102 | 59 | 13
  Grade 3 or Higher TEAE Related to Study Drug | 26 | 13 | 5
  Serious TEAE Related to Study Drug | 14 | 7 | 3

ADVERSE EVENTS:
Time Frame: All cause mortality: From the date of randomization up to 123 months and 24 days AE: From first dose on Day 1 until 28 days after the last dose of study drug, or one day before the date of initiation of cytotoxic chemotherapy or an investigational agent for treatment of prostate cancer, whichever comes first, up to 123 months and 24 days
Description: Data reported for deaths are the number of participants who died regardless of time (could be beyond treatment emergent adverse event time frame).
Groups:
- Placebo: Participants received enzalutamide matching placebo orally once a day during DB period until PSA progression and radiographic disease progression were centrally confirmed and 1 of the following 2 events became applicable to the participants: (1) initiation of cytotoxic chemotherapy or (2) initiation of an investigational agent for treatment of prostate cancer (up to 18.6 months).
- Placebo Patients Crossover to Enzalutamide 160 mg: Eligible participants who received enzalutamide matching placebo during DB period and who provided consent to take part in OLP, received 160 mg of enzalutamide orally once a day during open-label period until PSA progression and radiographic disease progression were centrally confirmed and 1 of the following 2 events became applicable to the participants: (1) initiation of cytotoxic chemotherapy or (2) initiation of an investigational agent for treatment of prostate cancer (up to 53.8 months).
Arm/Group | Enzalutamide | Placebo | Placebo Patients Crossover to Enzalutamide 160 mg
All-Cause Mortality (participants affected / at risk) | 85/202 | 57/193 | 21/51
Serious Adverse Events (participants affected / at risk) | 87/202 | 57/193 | 24/51
Other Adverse Events (participants affected / at risk) | 169/202 | 125/193 | 31/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzalutamide (N=202) | Placebo (N=193) | Placebo Patients Crossover to Enzalutamide 160 mg (N=51)
Anaemia (Blood and lymphatic system disorders) | 4 (6) | 4 (4) | 1 (1)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 5 (5) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0)
Angle closure glaucoma (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 2 (2) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric mucosal lesion (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Asthenia (General disorders) | 3 (3) | 2 (3) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 2 (2) | 3 (3) | 1 (1)
Disease progression (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hernia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Arthritis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Chronic sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Helicobacter infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Large intestine infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 16 (17) | 0 (0) | 3 (3)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 2 (2) | 1 (1) | 2 (3)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (2) | 1 (1) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (3)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Prostatic specific antigen increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (2)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (3) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (5) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Malignant neoplasm of thorax (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastases to bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Metastases to rectum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 0 (0) | 0 (0)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (3) | 0 (0)
Spinal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Cerebral thrombosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Cerebrovascular insufficiency (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 3 (4) | 0 (0) | 1 (2)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Myelopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Nerve compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Organic brain syndrome (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 4 (6) | 1 (1) | 1 (1)
Azotaemia (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 2 (3) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 8 (10) | 6 (6) | 0 (0)
Haemorrhage urinary tract (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 3 (3) | 1 (1) | 2 (2)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Ureteric rupture (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 7 (7) | 2 (2) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Prostatic haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Bilateral orchidectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Chemotherapy (Surgical and medical procedures) | 1 (1) | 4 (4) | 0 (0)
Medical device change (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Nephrostomy tube removal (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Radiotherapy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Spinal laminectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Tumour excision (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Ureteral stent insertion (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Ureteral stent removal (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 3 (4) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Malignant hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 1 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzalutamide (N=202) | Placebo (N=193) | Placebo Patients Crossover to Enzalutamide 160 mg (N=51)
Anaemia (Blood and lymphatic system disorders) | 30 (45) | 16 (25) | 10 (13)
Constipation (Gastrointestinal disorders) | 27 (31) | 15 (15) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 8 (12) | 4 (5) | 4 (6)
Nausea (Gastrointestinal disorders) | 23 (32) | 11 (12) | 2 (2)
Vomiting (Gastrointestinal disorders) | 11 (11) | 7 (8) | 0 (0)
Asthenia (General disorders) | 11 (13) | 7 (7) | 2 (2)
Fatigue (General disorders) | 29 (36) | 15 (20) | 3 (4)
Oedema peripheral (General disorders) | 14 (20) | 6 (8) | 4 (7)
Pyrexia (General disorders) | 12 (13) | 11 (14) | 0 (0)
Nasopharyngitis (Infections and infestations) | 22 (28) | 7 (7) | 3 (3)
Periodontitis (Infections and infestations) | 5 (12) | 1 (1) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 13 (19) | 5 (5) | 6 (6)
Weight decreased (Investigations) | 23 (28) | 11 (14) | 5 (8)
Decreased appetite (Metabolism and nutrition disorders) | 37 (52) | 19 (20) | 6 (6)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (10) | 1 (3) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 26 (32) | 12 (17) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 37 (48) | 19 (23) | 5 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 19 (28) | 24 (29) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 14 (16) | 5 (6) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 24 (31) | 17 (20) | 0 (0)
Dizziness (Nervous system disorders) | 22 (24) | 8 (8) | 4 (4)
Insomnia (Psychiatric disorders) | 18 (20) | 5 (5) | 0 (0)
Dysuria (Renal and urinary disorders) | 17 (19) | 7 (9) | 1 (2)
Haematuria (Renal and urinary disorders) | 12 (14) | 11 (14) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 14 (17) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 7 (7) | 5 (8)
Hypertension (Vascular disorders) | 21 (32) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data or 18 months after study completion date at all sites, whichever is first. Sponsor must receive a site's manuscript at least 45 days prior to publication for review and comment. If requested Sponsor may delay the publication for up to 60 days to seek patent protection.